CLINICAL TRIAL: NCT05389020
Title: Immunisation Simulation Using the Real-size Infant Manikin in Medical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Hartono Gunardi, MD, PhD, Prof, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 653/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2022-05-10; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Immunization Skills
Keywords: Simulation; Manikin; Immunization; Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 70 minutes course using newly developed real-size infant's arm and leg manikin
  Interventions: Other: Newly developed real-size infant's arm and leg manikin
- Control group (No Intervention): 70 minutes course using conventional manikin

INTERVENTIONS:
Other: Newly developed real-size infant's arm and leg manikin — The control group used conventional manikins made by Nasco; meanwhile, two newly designed real-size manikins were prepared for the intervention group: the right arm and right leg. Real-size manikins were developed based on the mean of anthropometric measurement of 50 Indonesian infants' arms and legs of healthy term neonates born in Dr Cipto Mangunkusumo Hospital. The manikins were made of Thermoplastic Polyurethane (TPU) filament using three-dimensional (3D) printing technology. The manufacturing process was carried out by the Medical Physics Department, Universitas Indonesia.
  Arms: Intervention group

SUMMARY:
This was a quasi-experimental study that comprised medical students in pediatric rotation at the Faculty of Medicine, Universitas Indonesia, Jakarta. The investigators determined students' knowledge and practice improvement through simulation by using the real-size infant's arm and leg manikins; and evaluate the confidence in immunization after the simulation.

ELIGIBILITY:
Inclusion Criteria:

* Medical students in paediatric rotation at the Faculty of Medicine, Universitas Indonesia, Jakarta
* Medical students who attended immunisation workshops

Exclusion Criteria:

* Students who refused to participate
* Students who did not attend the immunisation workshops

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Knowledge pre- and post-test questionnaire | Seven weeks after the immunization course
  The improvement of students' knowledge by using the real-size infant's arm and leg manikins
Practical skill score using rubric | Seven weeks after the immunization course
  The improvement of students' practical skill by using the real-size infant's arm and leg manikins
Number of students who were confident by self assessment using Likert scale questionnaire | Seven weeks after the immunization course
  The confidence in doing the immunization practice after the workshop
Students' feedback questionnaire | Seven weeks after the immunization course
  Students' response and feedback regarding the practice using the real-size infant's arm and leg manikins

CONTACTS AND LOCATIONS:
Overall Officials: Hartono Gunardi, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Indonesia